CLINICAL TRIAL: NCT05791097
Title: AdvanTIG-306: A Randomized, Double-blind, Placebo-controlled, Phase III Study Evaluating the Efficacy and Safety of Ociperlimab (WCD118/BGB-A1217) Combined With Tislelizumab (VDT482/BGB-A317) Plus Platinum-based Doublet Chemotherapy Versus Placebo Combined With Pembrolizumab Plus Platinum-based Doublet Chemotherapy as First-line Therapy for Participants With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study of Efficacy and Safety of Ociperlimab in Combination With Tislelizumab and Platinum-based Doublet Chemotherapy as First-line Treatment for Participants With Locally Advanced or Metastatic NSCLC.
Acronym: AdvanTIG-306
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision, not driven by safety concerns; no new safety signals have been observed in the ociperlimab program.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CWCD118A12301; 2022-503098-12-00 (Other: EU CTIS number)
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: AdvanTIG-306; ociperlimab; tislelizumab; pembrolizumab; carboplatin; cisplatin; paclitaxel; nab-paclitaxel; pemetrexed; squamous; non-squamous; non-small cell lung cancer; NSCLC; PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; pembrolizumab; Carboplatin; Cisplatin; Pemetrexed; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Ociperlimab + tislelizumab + chemotherapy (Experimental): Participants will receive ociperlimab in combination with tislelizumab and platinum-based doublet chemotherapy
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Arm B: Placebo + pembrolizumab + chemotherapy (Active Comparator): Participants will receive ociperlimab placebo in combination with pembrolizumab and platinum-based doublet chemotherapy
  Interventions: Drug: Placebo; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Arm C: Placebo + tislelizumab + chemotherapy (Placebo Comparator): Participants will receive ociperlimab placebo in combination with tislelizumab and platinum-based doublet chemotherapy
  Interventions: Drug: Placebo; Drug: Tislelizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Ociperlimab — Ociperlimab is a monoclonal antibody formulated for intravenous infusion. 900 mg of ociperlimab will be administered on Day 1 of each 21-day cycle
  Other Names: WCD118
  Arms: Arm A: Ociperlimab + tislelizumab + chemotherapy
Drug: Placebo — Placebo infusions will consist of a sterile, normal saline solution. Placebo will be administered on Day 1 of each 21-day cycle
  Arms: Arm B: Placebo + pembrolizumab + chemotherapy; Arm C: Placebo + tislelizumab + chemotherapy
Drug: Tislelizumab — Tislelizumab is a monoclonal antibody formulated for intravenous infusion. 200 mg of tislelizumab will be administered on Day 1 of each 21-day cycle
  Other Names: VDT482
  Arms: Arm A: Ociperlimab + tislelizumab + chemotherapy; Arm C: Placebo + tislelizumab + chemotherapy
Drug: Pembrolizumab — Pembrolizumab is a monoclonal antibody formulated for intravenous infusion. 200 mg of pembrolizumab will be administered on Day 1 of each 21-day cycle
  Arms: Arm B: Placebo + pembrolizumab + chemotherapy
Drug: Carboplatin — Carboplatin is a chemotherapy agent formulated for intravenous infusion. Carboplatin will be administered (AUC 6 mg/mL*min) on Day 1 of each 21-day cycle
Drug: Cisplatin — Cisplatin is a chemotherapy agent formulated for intravenous infusion. Cisplatin will be administered (75 mg/m^2) on Day 1 of each 21-day cycle
Drug: Pemetrexed — Pemetrexed is a chemotherapy agent formulated for intravenous infusion. Pemetrexed will be administered (500 mg/m^2) on Day 1 of each 21-day cycle
Drug: Paclitaxel — Paclitaxel is a chemotherapy agent formulated for intravenous infusion. Paclitaxel will be administered (200 mg/m^2) on Day 1 of each 21-day cycle
Drug: Nab-paclitaxel — Nab-paclitaxel is a chemotherapy agent formulated for intravenous infusion. Nab-paclitaxel will be administered (100 mg/m^2) on Day 1, 8 and 15 of each 21-day cycle

SUMMARY:
The primary scientific question of interest is whether the addition of ociperlimab to platinum-based chemotherapy and tislelizumab improve progression-free survival (PFS) or overall survival (OS) compared to pembrolizumab and platinum-based chemotherapy as first-line therapy for participants with locally advanced or metastatic squamous or non-squamous NSCLC with PD-L1 expression of ≥1%.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, multicenter, phase III study evaluating the efficacy and safety of ociperlimab in combination with tislelizumab and platinum-based doublet chemotherapy as first-line treatment for participants with locally advanced or metastatic NSCLC without actionable driver mutations.

Participants will receive study treatment every three weeks and will continue to receive it until RECIST 1.1 disease progression as determined by Investigator and confirmed by BIRC, unacceptable toxicity that precludes further treatment, treatment is discontinued at the discretion of the Investigator or participant, participant withdrawal of consent, pregnancy, lost to follow-up, or death.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed locally advanced (stage IIIb/IIIc not eligible for definitive chemoradiation, radiation or surgery) or metastatic (stage IV) NSCLC (according to AJCC: Cancer Staging Manual, 8th edition) participants with no previous systemic treatment for advanced disease.
* Known PD-L1 status determined, prior to study randomization
* At least one measurable lesion as defined by RECIST 1.1 according to local radiology assessment at screening.
* ECOG performance status ≤1.

Key Exclusion Criteria:

* Active autoimmune diseases requiring treatment with steroids or immunosuppressors in the past 2 years prior to randomization.
* History of severe hypersensitivity reaction or any contraindication to ociperlimab, tislelizumab, pembrolizumab (or any other monoclonal antibodies), platinum containing drugs, nab-paclitaxel, paclitaxel, pemetrexed or any known excipients of these drugs.
* Participants with known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Participants with documented epidermal growth factor receptor (EGFR) sensitizing mutations, and/or ALK rearrangement assessed as part of the patients's standard of care by a validated test, as per local regulations will be excluded from the study.
* Participants with other known druggable molecular drivers (any histology) such as BRAF V600, KRASG12C, MET exon 14 mutations, NTRK, RET or ROS-1 rearrangement diagnosed per local tests who might be candidates for alternative targeted therapies as applicable per local regulations and treatment guidelines are excluded.

Other inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-28 (Estimated); Primary Completion 2027-12-24 (Estimated); Study Completion 2027-12-26 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) based on Blinded Independent Review Committee (BIRC) assessment as per RECIST 1.1 in participants with PD-L1 expression in ≥1% of tumor cells (Arm A and B) | Up to 30 months
  Time from date of randomization/start of treatment to the date of event defined as the first documented progression based on BIRC assessment as per RECIST 1.1 or death due to any cause in participants with PD-L1 expression in ≥1% of tumor cells, for participants in Arm A compared to Arm B
Overall survival (OS) in participants with PD-L1 expression in ≥1% of tumor cells (Arm A and B) | Up to 52 months
  Time from date of randomization/start of treatment to date of death due to any cause in participants with PD-L1 expression in ≥1% of tumor cells, for participants in Arm A compared to Arm B

SECONDARY OUTCOMES:
PFS based on BIRC assessment as per RECIST 1.1 in all participants regardless of PD-L1 status (Arm A and B) | Up to 30 months
  Time from date of randomization/start of treatment to the date of event defined as the first documented progression based on BIRC assessment as per RECIST 1.1 or death due to any cause in all participants in Arm A compared to Arm B
OS in all participants regardless of PD-L1 status (Arm A and B) | Up to 52 months
  Time from date of randomization/start of treatment to date of death due to any cause in all participants in Arm A compared to Arm B.
Overall response rate (ORR) based in BIRC assessment as per RECIST 1.1 (Arm A and B) | Up to 30 months
  Percentage of participants with best overall response of complete response (CR) or partial response (PR) based in BIRC assessment as per RECIST 1.1 in participants with PD-L1 expression ≥1% and in all participants randomized, for participants in Arm A compared to Arm B
Disease Control Rate (DCR) based in BIRC assessment as per RECIST 1.1 (Arm A and B) | Up to 30 months
  Percentage of participants with best overall response of CR, PR or stable disease (SD)based in BIRC assessment as per RECIST 1.1 in participants with PD-L1 expression ≥1% and in all participants randomized, for participants in Arm A compared to Arm B
Time to response (TTR) based in BIRC assessment as per RECIST 1.1 (Arm A and B) | Up to 30 months
  Time from the date of randomization to the date of first documented response (CR or PR) based in BIRC assessment as per RECIST 1.1 in participants with PD-L1 expression ≥1% and in all participants randomized, for participants in Arm A compared to Arm B
Duration of response (DOR) based in BIRC assessment as per RECIST 1.1 (Arm A and B) | Up to 30 months
  Time between the date of first documented response (CR or PR) and the date of first documented progression or death due to any cause based in BIRC assessment as per RECIST 1.1 in participants with PD-L1 expression ≥1% and in all participants randomized, for participants in Arm A compared to Arm B
ORR based in BIRC assessment as per RECIST 1.1 (Arm A and C) | Up to 30 months
  Percentage of participants with best overall response of complete response (CR) or partial response (PR) based in BIRC assessment as per RECIST 1.1 in participants with PD-L1 expression ≥1% and in all participants randomized, for participants in Arm A compared to Arm C
DCR based in BIRC assessment as per RECIST 1.1 (Arm A and C) | Up to 30 months
  Percentage of participants with best overall response of CR, PR or stable disease (SD)based in BIRC assessment as per RECIST 1.1 in participants with PD-L1 expression ≥1% and in all participants randomized, for participants in Arm A compared to Arm C
TTR based in BIRC assessment as per RECIST 1.1 (Arm A and C) | Up to 30 months
  Time from the date of randomization to the date of first documented response (CR or PR) based in BIRC assessment as per RECIST 1.1 in participants with PD-L1 expression ≥1% and in all participants randomized, for participants in Arm A compared to Arm C
DOR based in BIRC assessment as per RECIST 1.1 (Arm A and C) | Up to 30 months
  Time between the date of first documented response (CR or PR) and the date of first documented progression or death due to any cause based in BIRC assessment as per RECIST 1.1 in participants with PD-L1 expression ≥1% and in all participants randomized, for participants in Arm A compared to Arm C
PFS based on BIRC assessment as per RECIST 1.1 (Arm A and C) | Up to 30 months
  Time from date of randomization/start of treatment to the date of event defined as the first documented progression based on BIRC assessment as per RECIST 1.1 or death due to any cause in participants with PD-L1 expression ≥1% and in all participants randomized, for participants in Arm A compared to Arm C
Pharmacokinetic (PK) parameter: Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of ociperlimab and tislelizumab | Up to 30 months
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of ociperlimab and tislelizumab. AUClast will be summarized using descriptive statistics.
PK parameter: Maximum concentration (Cmax) of ociperlimab and tislelizumab | Up to 30 months
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of ociperlimab and tislelizumab. Cmax will be summarized using descriptive statistics.
PK parameter: Time to reach maximum concentration (Tmax) of ociperlimab and tislelizumab | Up to 30 months
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of ociperlimab and tislelizumab. Tmax will be summarized using descriptive statistics.
PK parameter: Lowest serum concentration reached before the next dose is administered (Ctrough) of ociperlimab and tislelizumab | Up to 30 months
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of ociperlimab and tislelizumab. Ctrough will be summarized using descriptive statistics.
PK parameter: AUC calculated at the end of the dosing interval (AUCtau)of ociperlimab and tislelizumab | Up to 30 months
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of ociperlimab and tislelizumab. AUCtau will be summarized using descriptive statistics.
Immunogenicity: Anti-drug antibodies (ADA) prevalence at baseline of ociperlimab and tislelizumab | Baseline
  Prevalence of ADA (anti-ociperlimab, anti-tislelizumab) at baseline is defined as the percentage of participants who have an ADA positive result at baseline
Immunogenicity: ADA incidence following treatment with ociperlimab and tislelizumab | Up to 30 months
  Incidence of ADA (anti-ociperlimab, anti-tislelizumab) on treatment is defined as the percentage of participants who are treatment-induced ADA positive (post-baseline ADA positive with ADA-negative sample at baseline) and treatment-boosted ADA positive (post-baseline ADA positive with titer that is at least the fold titer change greater than the ADA-positive baseline titer)
Time to definitive 10-point deterioration in physical and role functioning on the EORTC QLQ-C30 questionnaire | Up to 30 months
  The EORTC QLQ-C30 is a questionnaire developed to assess the health-related quality of life of cancer participants. It assesses 15 domains consisting of 5 functional domains (physical, role, emotional, cognitive, social) and 9 symptom domains (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties) and a global health status/quality of life (QoL) scale. All of the domain scores range from 0 to 100. A high score for a functional scale indicates a high and healthy level of functioning but a high score for a symptom scale indicates a high level of symptoms.
  The time to definitive 10 point deterioration of physical functioning and role functioning is defined as the time from the date of randomization to first onset of ≥10 points increase from baseline (worsening) of the corresponding scale score, with no later change below this threshold or death due to any cause.
Time to definitive 10-point deterioration in symptom scores for chest pain, cough and dyspnea on the EORTC QLQ-LC13 questionnaire | Up to 30 months
  The Lung Cancer module of the EORTC's quality of life questionnaire (EORTC QLQ-LC13) is used in conjunction with the EORTC QLQ-C30 and provides information on an additional 13 items specifically related to lung cancer. The lung cancer module incorporates one multi-item scale to assess dyspnea, and 9 single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All of the domain scores range from 0 to 100. A high score indicates a high level of symptoms.
  The time to first 10 point deterioration symptom scores of chest pain, cough and dyspnea is defined as the time from the date of randomization to first onset of ≥10 points increase from baseline (worsening) of the corresponding scale score, with no later change below this threshold or death due to any cause.
Time to confirmed 10-point deterioration in physical and role functioning on the EORTC QLQ-C30 questionnaire | Up to 30 months
  The EORTC QLQ-C30 is a questionnaire developed to assess the health-related quality of life of cancer participants. It assesses 15 domains consisting of 5 functional domains (physical, role, emotional, cognitive, social) and 9 symptom domains (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties) and a global health status/quality of life (QoL) scale. All of the domain scores range from 0 to 100. A high score for a functional scale indicates a high and healthy level of functioning but a high score for a symptom scale indicates a high level of symptoms.
  The time to confirmed 10-point deterioration of physical functioning and role functioning is defined as the time from the date of randomization to first onset of≥10 points deterioration from baseline and confirmed by a second consecutive ≥10 points deterioration from baseline, or one assessment followed by death from any cause before the next scheduled data collection.
Time to confirmed 10-point deterioration in symptom scores for chest pain, cough and dyspnea on the EORTC QLQ-LC13 questionnaire | Up to 30 months
  The Lung Cancer module of the EORTC's quality of life questionnaire (EORTC QLQ-LC13) is used in conjunction with the EORTC QLQ-C30 and provides information on an additional 13 items specifically related to lung cancer. The lung cancer module incorporates one multi-item scale to assess dyspnea, and 9 single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All of the domain scores range from 0 to 100. A high score indicates a high level of symptoms.
  The time to first 10 point deterioration symptom scores of chest pain, cough and dyspnea is defined as the time from the date of randomization to first onset of≥10 points deterioration from baseline and confirmed by a second consecutive ≥10 points deterioration from baseline, or one assessment followed by death from any cause before the next scheduled data collection.
Time to definitive 10-point deterioration in global health status/quality of life, shortness of breath and pain on the EORTC QLQ-C30 questionnaire | Up to 30 months
  The EORTC QLQ-C30 is a questionnaire developed to assess the health-related quality of life of cancer participants. It assesses 15 domains consisting of 5 functional domains (physical, role, emotional, cognitive, social) and 9 symptom domains (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties) and a global health status/quality of life (QoL) scale. All of the domain scores range from 0 to 100. A high score for a functional scale indicates a high and healthy level of functioning but a high score for a symptom scale indicates a high level of symptoms.
  The time to definitive 10-point deterioration in global health status/quality of life, shortness of breath and pain scores is defined as the time from the date of randomization to first onset of ≥10 points increase from baseline (worsening) of the corresponding scale score, with no later change below this threshold or death due to any cause.
Utility scores of the EQ-5D-5L | Up to 30 months
  EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.
Progression-free survival deferred (PFS2) | Up to 30 months
  Time from date of randomization to the first documented progression on next line therapy or death from any cause, whichever occurs first
Time to definitive deterioration of the ECOG performance status | Up to 30 months
  Time to definitive deterioration of the ECOG PS by one category of the score. The ECOG PS is a measure of functional status. It ranges from 0 to 5, with 0 denoting perfect health and 5 death. A deterioration is considered definitive if no improvements in the ECOG PS status is observed at any subsequent time of measurement during the treatment period following the time point where the deterioration is observed.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com